CLINICAL TRIAL: NCT02204059
Title: A Phase I Biodistribution Study With 186 Re-labelled Humanised Monoclonal Antibody BIWA 4, in Patients With Non-small Cell Lung Cancer
Brief Title: Biodistribution Study With 186 Re-labelled Humanised Monoclonal Antibody BIWA 4 in Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1170.3
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

ARMS (1):
- hMAb BIWA 4 (Experimental): Bivatuzumab: 186 Re-labelled humanised monoclonal antibody BIWA 4
  Interventions: Drug: hMAb BIWA 4

INTERVENTIONS:
Drug: hMAb BIWA 4

SUMMARY:
The primary objectives of this study is to assess the safety and tolerability of intravenously (i.v.) administered 186 Rhenium-isotope (186Re)-labelled bivatuzumab and to investigate the biodistribution and pharmacokinetics of 186 Re-labelled bivatuzumab in patients with non-small cell lung cancer (NSCLC)

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or cytological confirmation of Non small cell lung cancer (NSCLC) stage I, II or IIIa according to the staging system of the American Joint Committee on Cancer (AJCC)
* Patients destined for resection of the tumour
* Patients over 18 years of age
* Patients younger than 80 years of age
* Patients who had given 'written informed consent'
* Patients with a life expectancy of at least 3 months
* Patients with a good performance status: Karnofsky > 60

Exclusion Criteria:

* Life-threatening infection, allergic diathesis, organ failure (bilirubin > 30µmol/l and/or creatinine > 150 µmol/l) or evidence of a recent myocardial infarction on Electrocardiogram (ECG) or unstable angina pectoris
* Pre-menopausal women (last menstruation <= 1 year prior to study start)

  * Not surgically sterile (hysterectomy, tubal ligation) and
  * Not practicing acceptable means of birth control, (or not planned to be continued throughout the study). Acceptable methods of birth control include oral, implantable or injectable contraceptives
* Women with a positive serum pregnancy test at baseline
* White blood cell count < 3000/mm³, granulocyte count < 1500/mm³ or platelet count < 100000/mm³. Details of prior chemotherapy and radiotherapy had to be known.
* Hematological disorders, congestive heart failure, bronchial asthma, alimentary or contact allergy, severe atopy or allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 1999-12; Primary Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 6 weeks post infusion
Number of patients with abnormal changes in laboratory parameters | up to 6 weeks post infusion
Number of patients with clinically significant changes in vital signs | up to 6 weeks post infusion
Presence of Human-Anti-Human-Antibody (HAHA) | up to 6 weeks post infusion
Biodistribution of 186Re-labelled hMAb BIWA 4 in tumour and normal tissue samples | up to 96 hours post infusion
  assessed by radioimmunoscintigraphy expressed as no, low, medium or high
Uptake of 186Re-labelled hMAb BIWA 4 in tumour and normal tissue samples | after surgery on day 8
  Biodistribution assessed from biopsy sample as percentage of the injected dose per kg tissue (%ID/kg)
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 6 weeks post infusion
Cmax (Maximum measured concentration of the analyte in plasma) | up to 6 weeks post infusion
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 6 weeks post infusion
t½ (Terminal half-life of the analyte in plasma) | up to 6 weeks post infusion
MRT (Mean residence time of the analyte in the body) | up to 6 weeks post infusion
Vss (Apparent volume of distribution under steady state conditions) | up to 6 weeks post infusion
Vz (Apparent volume of distribution during the terminal phase) | up to 6 weeks post infusion
CL (Total body clearance) | up to 6 weeks post infusion